CLINICAL TRIAL: NCT04024449
Title: Colyak Hastaliginin Puberte ve Sonrasinda Over Fonksiyonlarina Etkisinin Arastirilmasi
Brief Title: Can Celiac Disease Affect Ovarian Function in Adolescent?
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018/166
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Celiac Disease; Ovarian Failure
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac Disease: Celiac disease with the following criteria;
  * 13 ≤ Age ≤20
  * At least one year after menarche
  * Non-obesity or malnutrition, Non-Hyperandogenism symptoms, and blood tests, Non-Hyper or hypothyroidism, Non-Hyperprolactinemia.
  Interventions: Other: Group A
- Control: The adolescent with the following criteria;
  * 13 ≤ Age ≤20
  * At least one year after menarche
  * Non-obesity or malnutrition, Non-Hyperandogenism symptoms, and blood tests, Non-Hyper or hypothyroidism, Non-Hyperprolactinemia.
  * Control group; with normal menstrual period, Non-chronic diseases
  Interventions: Other: Group A

INTERVENTIONS:
Other: Group A — ovarian function test in control group
  Other Names: Celiac disease

SUMMARY:
This case-control multicentre trial was performed from January 1, 2017, to May 31, 2018, in University of Health Sciences Bakirkoy Dr. Sadi Konuk Training and Research Hospital and Hitit University Hospital. Adolescents who were in compliance with the inclusion criteria were called by telephone for blood collection and ultrasound on the 3rd day of menstruation after approval from local ethical registration. On days 2-5 of the menstrual cycle, level of follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), prolactin (PRL), and AMH were measured from venous blood samples in both groups. Antral Follicle Counts (AFCs) and ovarian volumes were determined on the same day.

DETAILED DESCRIPTION:
This case-control multicentre trial was performed from January 1, 2017, to May 31, 2018, in University of Health Sciences Bakirkoy Dr. Sadi Konuk Training and Research Hospital and Hitit University Hospital. This study was conducted with approval from the BTRH ethical board (number: 2018/166). This study covered 20 cases suffered from Celiac Disease and 18 were with regular menstrual period and healthy adolescent girls. Adolescents who were in compliance with the inclusion criteria were called by telephone for blood collection and ultrasound on the 3rd day of menstruation after approval from local ethical registration. Data on age, body mass index (BMI), levels of antitransglutaminase immune globulins A (IgA), positivity to antiendomysium IgA were recorded. On days 2-5 of the menstrual cycle, level of follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), prolactin (PRL), and AMH were measured from venous blood samples in both groups. The samples were centrifuged at 3,000 rpm for 10 minutes to aliquot the supernatants. Antral Follicle Counts (AFCs) and ovarian volumes were determined on the same day by the same ultrasound devices. The inclusion criteria included the following items;

* 13 ≤ Age ≤20
* At least one year after menarche
* Non-obesity or malnutrition, Non-Hyperandogenism symptoms, and blood tests, Non-Hyper or hypothyroidism, Non-Hyperprolactinemia.
* Control group; with a normal menstrual period, Non-chronic diseases The study had exclusion criteria such as delayed menarche, early puberty, delayed puberty, delayed development of secondary sexual characters due to another sexual disorder.

IBM SPSS version 22.0 (IBM Corp., Armonk, NY, USA) was used for all data analyses. Descriptive statistics are presented as numbers and percentages (%) for qualitative variables and as mean ± standard deviation and median (range) for quantitative variables. Normality distribution of data was evaluated using Kolmogorov-Smirnov, and Shapiro-Wilk tests to guide statistical test choice.

ELIGIBILITY:
Inclusion Criteria:

* •Celiac disease and control group with 13 ≤ Age ≤20

  * At least one year after menarche

Exclusion Criteria:

* delayed menarche, early puberty, delayed puberty, delayed development of secondary sexual characters due to another sexual disorder, obesity or malnutrition, Hyperandrogenism symptoms, and blood tests, Hyper or hypothyroidism, Hyperprolactinemia.

Ages: 13 Years to 20 Years | Sex: Female
Age Groups: Child, Adult
Study Population: The study population included 37 subjects in total. 20 people were in patients with celiac disease, 17 people were healthy adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Anti mullerian Hormone (AMH) | on Day 3 menstruation
  Level of AMH
Follicle Situmulating Hormone (FSH) | on Day 3 menstruation
  Level of FSH
Ovarian Volume | on Day 3 menstruation
  Ovarian volume measurement via Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Atakan Comba, M.D., Study Chair — Hitit University Department of Pediatric Gastroenterology
Locations (1):
- Cihan Comba, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If the data is wanted, we will share data at any time.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Comba C, Comba A, Yilmaz H, Erdogan SV, Demir O. Celiac disease does not influence markers of ovarian reserve in adolescent girls. Arch Gynecol Obstet. 2020 Nov;302(5):1263-1269. doi: 10.1007/s00404-020-05666-4. Epub 2020 Jun 27. PMID 32594297